CLINICAL TRIAL: NCT05137483
Title: Comparison of Upper Extremity Functional Capacity, Respiratory Functions, Fatigue and Quality of Life in Chronic Obstructive Pulmonary Patients With and Without Cognitive Impairment
Brief Title: Cognitive Impairment and Upper Extremity Performance in COPD
Acronym: COPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof, Izmir Katip Celebi University
Other Study IDs: IKC125
Record Dates: First submitted 2021-11-18; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: COPD; Upper Extremity; Upper Limb Function; Cognitive Impairment
Keywords: copd; cognitive impairment; cognition; upper extremity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With cognitive impairment: Pulmonary function test, COPD assessment scale, Mini-Mental State Examination and Montreal Cognitive Assessment Scale, 6 min pegboard ring test, grip strength measurement, Fatigue Impact Scale and St.George Respiratory Questionnaire will be applied to the group.
  Interventions: Other: Functional tests
- without cognitive impairment: Pulmonary function test, COPD assessment scale, Mini-Mental State Examination and Montreal Cognitive Assessment Scale, 6 min pegboard ring test, grip strength measurement, Fatigue Impact Scale and St.George Respiratory Questionnaire will be applied to the group.
  Interventions: Other: Functional tests

INTERVENTIONS:
Other: Functional tests — We will apply upper extremity performance tests, hand grip measurements, and scales measuring fatigue and quality of life to the groups.

SUMMARY:
Within the scope of this study, COPD patients will be divided into two groups according to cognitive dysfunction.

Pulmonary function test, COPD assessment scale, Mini-Mental State Examination and Montreal Cognitive Assessment Scale, 6 min pegboard ring test, grip strength measurement, Fatigue Impact Scale and St.George Respiratory Questionnaire will be applied to the groups.

DETAILED DESCRIPTION:
Although the mechanism of cognitive dysfunction in COPD is not clear, the reasons focused on are; decreased oxygen use, high carbon dioxide levels, increased inflammation and oxidative stress, decreased physical activity, peripheral vascular diseases, atherosclerosis, high or low blood pressure, cerebral vasoconstriction, increased intracranial pressure, accompanying comorbidities, smoking and genetic predisposition, brain damage and exacerbations have been reported. Few studies have shown that cognitive dysfunction is associated with functional performance. There are no studies on the effect of cognitive function on upper extremity performance and mechanisms of action in COPD patients.

The aim of this study is to compare upper extremity functional capacities, respiratory functions, fatigue and quality of life in COPD patients with and without cognitive function impairment.

Within the scope of this study, COPD patients will be divided into two groups according to cognitive dysfunction.

Pulmonary function test, COPD assessment scale, Mini-Mental State Examination and Montreal Cognitive Assessment Scale, 6 min pegboard ring test, grip strength measurement, Fatigue Impact Scale and St.George Respiratory Questionnaire will be applied to the groups.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Stage 2-3-4 according to the GOLD classification in the 40-65 age range

Exclusion Criteria:

* Exacerbation of respiratory symptoms in the past 4 weeks (change in breathlessness and/or sputum volume/color, need for antibiotic treatment or need for hospitalization)
* Presence of asthma, unstable coronary heart disease, uncontrolled diabetes, hypertension, left-sided congestive heart failure, neoplasia, severe claudication, encephalitis or epilepsy
* Having a history of head trauma or brain tumor
* Having a significant psychiatric condition or the presence of defined dementia, according to the American Psychiatric Association

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COPD patients above 45 years
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-11-19 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
6 min. pegboard ring test | 6 minutes
  It is used to measure upper extremity functional capacity.

SECONDARY OUTCOMES:
Mini Mental State Test | 15 minutes
  It is used for measuring cognitive impairment
Montreal Cognitive Assessment Scale | 30 minutes
  It is used for measuring cognitive impairment
Respiratory Function Test | 20 minutes
  It is used for measuring lung functions and respiratory muscle strength
Fatigue Impact Scale | Time Frame: 20 minutes
  It is used for measuring fatigue level
St. George Respiratory Questionnaire | 20 minutes
  It is used for measuring desase-related quality of life
COPD Assessment Test | 10 minutes
  It is used for measuring health status of COPD patients
mMRC Dyspnea Scale | 5 minutes
  It is used for measuring dyspnea sensation in daily living activities

IPD SHARING:
Plan to Share IPD: No